CLINICAL TRIAL: NCT04154202
Title: The Role of NM/CT 870 DR Camera in the Diagnosis of Joint Prosthesis and Tibial Open Reduction and Internal Fixation (ORIF) Complications.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC-19-ES-0468-CTIL
Record Dates: First submitted 2019-10-29; First posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Bone Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bone inaction patients (Experimental): Three months or more post joint replacement, or post tibial ORIF, or last surgical intervention adult patients suspected of bone infection and or mechanical loosening.
  Interventions: Other: Bone Scan

INTERVENTIONS:
Other: Bone Scan — Bone Scan: three-phase planar Bone Scan and a SPECT/CT [perfusion, blood pool and SPECT/CT of the relevant region of interest (ROI), and a whole-body planar late bone scan].

SUMMARY:
This is a prospective study. Patients' cohort is composed of 70 consecutive post joint replacement and post tibial ORIF patients, referred by their orthopedic surgeon to the Nuclear Medicine institute of Tel Aviv Sourasky Medical Center in the diagnostic work up of post operative bone infection and or mechanical loosening.

The proposed study will be presented to the ethical committee of the medical center and will be started once approved.

ELIGIBILITY:
Inclusion Criteria:

1. Three months or more post joint replacement, or post tibial ORIF, or last surgical intervention adult patients suspected of bone infection and or mechanical loosening.

Exclusion Criteria:

1. Patients younger than 18 years;
2. Shorter than 3 month surgical intervention at the suspected area; Newly diagnosed (<3 months) fractures around the prosthesis;
3. Pathological fractures (e.g. Metastatic).

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-11-15 (Estimated); Primary Completion 2020-01-15 (Estimated); Study Completion 2021-11-15 (Estimated)

PRIMARY OUTCOMES:
To assess the role of NM imaging in the diagnosis work up of joint prosthesis and tibial ORIF complications by using GE NM/CT 870 DR camera and its accompanied tools.. | 1 year

IPD SHARING:
Plan to Share IPD: Undecided